CLINICAL TRIAL: NCT05076955
Title: Evaluating the Healing of Diabetic Foot Ulcers With Compounded Anti-Infective Irrigation
Brief Title: Evaluating the Healing of Diabetic Foot Ulcers With Compounded Anti-Infective Irrigation Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Keystone Pharmacy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-UMC014
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of Diabetic Foot Ulcer (Experimental): Participants with diabetic foot ulcers will be treated with a compounded, anti-infective irrigation therapy daily until closure of the ulcer or up to a maximum of 3 months. This is an irrigating foot bath with a compounded medication of vancomycin-tobramycin-itraconazole. This medication with combined 3/4 gallon of water. Participant will soak foot in solution for 10 minutes per day. Daily until wound is healed for a minimum of 4 weeks and a maximum of 3 months.
  Interventions: Drug: vancomycin-tobramycin-itraconazole

INTERVENTIONS:
Drug: vancomycin-tobramycin-itraconazole — Participants with diabetic foot ulcers will be treated with a compounded, anti-infective irrigation therapy daily until closure of the ulcer or up to a maximum of 3 months. This is an irrigating foot bath with a compounded medication of vancomycin-tobramycin-itraconazole. This medication with combined 3/4 gallon of water. Participant will soak foot in solution for 10 minutes per day. Daily until wound is healed for a minimum of 4 weeks and a maximum of 3 months.

SUMMARY:
Diabetic foot ulcers (DFUs) are a frequent clinical problem observed in diabetic patients. Properly managed, most can be cured, but many patients needlessly undergo amputations because of improper diagnostic and therapeutic approaches. The purpose of this study is to evaluate the effectiveness of a compounded, anti-infective irrigation therapy to increase the healing rates of diabetic foot ulcers and thereby provide a new therapeutic option for health care providers treating high-risk patients with DFUs regardless if secondary fungal infections are present.

Participants diagnosed with diabetes type 1 or 2 and with a documented open diabetic foot ulcer/wound with or without a secondary fungal infection will be included in this prospective, active intervention pilot study. Healing rates will be evaluated every two weeks following the initiation of study therapy up to three months. Participants with diabetic foot ulcers will be treated with a compounded, anti-infective irrigation therapy daily until closure of the ulcer or up to a maximum of 3 months. Participants will be asked to return to clinic every two - four weeks for assessment of the ulcer and compliance with treatment.

A sample size of approximately 100 patients is estimated to have 90% power to detect 15% improvement in ulcer healing rates to 45% and 35% compared to historical benchmarks of approximately 30% for ulcers of <6 months duration and 20% for ulcers ≥6 months duration and/or prior treatment failure, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* An open DFU / wound of any size (including those requiring debridement in operation room or clinic setting) with or without a secondary fungal infection
* ≥ 18 years of age
* Treatment naïve or treatment failure with oral antibiotics to current wound infection

Exclusion Criteria:

* Patients who present with untreated or on active-treatment for osteomyelitis, exposed bone, or have a life-threatening need of immediate surgery.
* Patients who are allergic to any components of the investigated product.
* Patients who have ≥ 15 shoe size
* Patients who have received IV antibiotics within the past 30 days
* Patients with HgbA1C > 14
* Patients on active cancer treatment
* Patients needing re-vascularization of the affected area but did not receive treatment.
* Patients diagnosed with HIV/AIDs
* Patients unable or unwilling to obtain and wear off-loading footwear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Healing Rate | 12 weeks
  We will be looking at measurements of the wound at the start of the study and at each study visit until the wound is healed, or the study has ended. The wounds are measured with a ruler by the provider seeing the patient at the time of the visit in centimeters. The wounds are also photographed with a ruler in the photograph for size.

SECONDARY OUTCOMES:
Wound Closure | Until the wound is closed up to 12 weeks
  Assessing how many patients wounds closed during the study and the time in weeks it took for the patient to close their wound.

CONTACTS AND LOCATIONS:
Overall Officials: Laura R Vick, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share deidentified data that is collected in the study in full. All IPD that will result in publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study for a period of 6 months or until publication.

REFERENCES:
- [Background] Lipsky BA, Berendt AR, Cornia PB, Pile JC, Peters EJ, Armstrong DG, Deery HG, Embil JM, Joseph WS, Karchmer AW, Pinzur MS, Senneville E; Infectious Diseases Society of America. 2012 Infectious Diseases Society of America clinical practice guideline for the diagnosis and treatment of diabetic foot infections. Clin Infect Dis. 2012 Jun;54(12):e132-73. doi: 10.1093/cid/cis346. PMID 22619242
- [Background] Everett E, Mathioudakis N. Update on management of diabetic foot ulcers. Ann N Y Acad Sci. 2018 Jan;1411(1):153-165. doi: 10.1111/nyas.13569. PMID 29377202